CLINICAL TRIAL: NCT01427764
Title: Dentin Hypersensitivity Following Non-surgical Periodontal Therapy With Hand or Ultrasonic Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: Principal Investigator, ERICA DEL PELOSO RIBEIRO, PhD in Periodontics, Escola Bahiana de Medicina e Saude Publica
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2011-08-24; First posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Periodontal Disease; Dentin Sensitivity
Keywords: Dentin sensitivity; Dental scaling; Ultrasonic; manual and ultrasonic instrumentation
MeSH Terms: conditions — Periodontal Diseases; Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Device: manual and ultrasonic instruments — The individuals were instructed regarding causes and consequences of periodontal disease as well as prevention techniques, including the sulcular brushing technique and flossing. The retention factors of plaque (caries cavities, excess supragingival restorations and calculus) were removed during the initial visits. Clinical parameters were initially assessed 30 days after initial therapy.
  The quadrants were randomly assigned and a total of 28 teeth were examined and treated. One side was treated with Gracey curettes (Hu-Friedy™ - Chicago, IL, USA) - control group and the other side with ultrasonic instruments (Profi II Ceramic™, Dabi Atlante - Ribeirão Preto, São Paulo, Brazil) - the test group, using the tip for subgingival instrumentation Perio Sub (Dabi Atlante ®).

SUMMARY:
Periodontal instrumentation aims to remove plaque and calculus from the root surface. Both manual and ultrasonic instruments have been used for such decontamination; however, establishing a healthy periodontium can result in adverse effects, such as dentin hypersensitivity. The aim of this study was to evaluate the effects of hand or ultrasonic instrumentation on dentin hypersensitivity in patients undergoing non-surgical periodontal treatment. For this controlled clinical trial of a "split mouth" design, 14 patients were selected with homologous teeth in the incisor to premolar region and probing depth ≥ 5 mm on the buccal aspect of the teeth. One side (control) was instrumented with hand instruments and the other side (test) with ultrasonic instruments. Dentin hypersensitivity was assessed in the baseline and during the follow 4 weeks after treatment, with a periodontal probe scratching the root surface and with an air jet. The patient's response was detected by a visual analog scale (VAS) of 10 cm.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with chronic or aggressive periodontitis, according to the American Academy of Periodontology classification15, requiring non-surgical periodontal treatment in at least two quadrants. These quadrants should present two contralateral and homologous teeth in the incisor to premolar region with probing depth ≥ 5 mm and bleeding on probing on the buccal surface.

Exclusion Criteria:

* presence of systemic illness or medication use (six months preceding the research), which could influence the response to periodontal treatment,
* performance of periodontal treatment including subgingival instrumentation in the six months preceding the study,
* performance of treatment for dentin hypersensitivity in the three months previous to the study,
* presence of periapical or pulpal changes,
* being under orthodontic treatment,
* smoking and
* pregnancy.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

SECONDARY OUTCOMES:
Change in the clinical attachment level | baseline and 4 weeks follow after treatment
  Measured by a calibrated professional on baseline and 30 days after treatment - the distance from the cemental enamel junction to the bottom of the pocket.